CLINICAL TRIAL: NCT06418269
Title: The Effect of Insulin Education Given to Children With Diabetes by Therapeutic Play Method on Anxiety and Fear Levels
Brief Title: The Effect of Therapeutic Play on Anxiety and Fear Levels in Children With Diabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Canan Genç, Research Assistant, Fenerbahce University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 53.2024fbu
Record Dates: First submitted 2024-05-13; First posted 2024-05-17 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-01

CONDITIONS: Type1diabetes; Therapeutic Play; Fear State; Anxiety State
Keywords: Type1diabetes; Therapeutic play; Fear state; Anxiety State
MeSH Terms: conditions — Anxiety Disorders | interventions — Play Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Therapeutic Play Group (Experimental)
  Interventions: Other: Therapeutic Play
- Control Group (No Intervention)

INTERVENTIONS:
Other: Therapeutic Play — Children will be asked to fill in the "Child Patient Identification Form", "State Anxiety Scale in Children" and "Child Fear Scale" 30 minutes before insulin treatment. Before the insulin treatment, the children in the experimental group will have their blood glucose measured and insulin administered on a doll using the therapeutic play method. The child will be told that the doll is hospitalized with a diagnosis of Type 1 diabetes and will be expected to assume the role of a nurse to administer insulin to the doll. Then, the steps of blood glucose measurement and insulin treatment (subcutaneous) will be explained to the child and the child will be asked to administer insulin to the baby. Within 10 minutes after subcutaneous insulin treatment, the child will be asked to fill out the "State Anxiety Scale in Children" and "Child Fear Scale".
  Arms: Therapeutic Play Group

SUMMARY:
The study will be conducted using a randomized controlled method. Children with type 1 diabetes who are admitted to the Pediatric Endocrinology Service will be divided into two groups by randomization method. Following randomization, children in the experimental group will play a therapeutic game before their subcutaneous insulin treatment. In the subcutaneous insulin treatment of the children in the control group, the routine practice of the clinic will be applied. Anxiety and fear levels of all children in the experimental and control groups will be evaluated before and after subcutaneous insulin treatment.

DETAILED DESCRIPTION:
Excessive stress and anxiety experienced by children can affect their physical and physiological health and hinder their ability to cope with medical interventions. Pain and negative emotions associated with blood sampling or insulin administration can negatively affect children's diabetes self-care skills and may lead to avoidance of injections.

Play-based interventions allow the child to process potentially frightening events and correct misconceptions about an illness and its management. Overall, therapeutic play interventions have been effective in reducing the child's pain, anxiety and stress while encouraging cooperation. Since insulin treatment (subcutaneous) causes fear and anxiety in children, the aim of this study was to reduce fear and anxiety by dramatization method by storytelling the child's procedure and disease with the game of administering insulin treatment (subcutaneous) to a doll.

In the Pediatric Endocrinology Service, children between the ages of 9 and 12 years who have just been diagnosed with Type 1 diabetes and who meet the sample selection criteria and their parents will be met and informed about the study and written and verbal consent will be obtained from the children and their parents who volunteer to participate in the study. Children will be asked to fill out the "Child Patient Identification Form", "State Anxiety Scale in Children" and "Child Fear Scale" 30 minutes before insulin treatment. Then, the children will be randomized by the researcher and assigned to two different groups as experimental and control groups. Before the insulin treatment procedure, the children in the experimental group will be made to take blood glucose and administer insulin on a doll with the therapeutic play method. The children in the control group will receive the routine treatment of the clinic. Within 10 minutes after subcutaneous insulin treatment, the child will be asked to fill out the "State Anxiety Scale in Children" and "Child Fear Scale".

Therapeutic Play Content: The doll to be used in the study represents the sick children in the experimental group. The child will be told that the doll has been hospitalized with a diagnosis of Type 1 diabetes and will be expected to assume the role of a nurse in order to administer insulin to the doll. The materials to be used during insulin administration will be introduced to the child and the child will be made to recognize the materials more closely. Then, the steps of blood glucose measurement and insulin treatment (subcutaneous) will be explained to the child and the child will be asked to apply the insulin to the doll.

ELIGIBILITY:
Inclusion Criteria:

* The child must be between the ages of 9 and 12 (since the State Anxiety Inventory for Children Scale is for this age range)
* Diagnosed with type 1 diabetes
* Absence of mental retardation
* Receiving subcutaneous insulin treatment for the first time
* Voluntariness of the child and parent to participate in the study

Exclusion Criteria:

* Visual, hearing or speech impairment
* Illiteracy of the child
* Having a clinical condition that prevents playing games (excessive fatigue, weakness, etc.)

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-07-18 (Estimated); Primary Completion 2026-06-18 (Estimated); Study Completion 2026-08-18 (Estimated)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory for Children | 30 minutes before insulin treatment, within 10 minutes after subcutaneous insulin treatment
  Anxiety states of children that may occur due to subcutaneous insulin treatment will be evaluated. The lowest score that can be obtained from the State Anxiety Scale is 20 and the highest score is 60.
Child Fear Scale | 30 minutes before insulin treatment, within 10 minutes after subcutaneous insulin treatment
  Fear states of children that may occur due to subcutaneous insulin treatment will be evaluated. In this method, the child is shown a picture with five facial expressions rated between 0 and 4. 0 indicates no fear and anxiety, while 4 indicates the highest fear and anxiety.

IPD SHARING:
Plan to Share IPD: No